CLINICAL TRIAL: NCT01935310
Title: Clinical and Histological Analysis of Photoaging Treatment With Imiquimod Cream 5%
Brief Title: Photoaging Treatment With Imiquimod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Sol Beatriz Jiménez, Researcher, CES University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IMQ003
Record Dates: First submitted 2013-08-14; First posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-08

CONDITIONS: Photoaging
Keywords: Photoaging; imiquimod; wrinkles; elastosis
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- imiquimod use in photoaging (Experimental): Evaluate the efficacy and safety of imiquimod as a treatment option for photoaging photoaging equal to or greater than 3.
  Interventions: Drug: Imiquimod

INTERVENTIONS:
Drug: Imiquimod — From the group of subjects who met the inclusion criteria, 22 people were selected randomly (using a random number table) since a 20-25% loss to follow up was calculated and the least amount of patients needed were 17.
  During the study participants applied imiquimod cream 5% (Virosupril ® laboratories Roemmers) in the periocular area during the night, three times a week, on nonconsecutive days, for 12 weeks (3 months). If patients presented irritative dermatitis a topical 0.05% desonide cream was administered and applied for less of 5 days until symptoms improved.
  Other Names: Virosupril®

SUMMARY:
Recently it was demonstrated that imiquimod in addition to exerting a repairing effect in pre malignant and malignant lesions caused by UV radiation it reverses histopathological changes associated with the photoaging skin.

This is an experimental exploratory study. It included 17 patients. The patients were diagnosed with photoaging grades III and IV in the scale of Glogau and volunteered to participate in the study. Patients were treated with imiquimod 5% topically, for a time period of 12 weeks. Biopsies were taken from periorbital skin area at baseline and after 4 weeks after completing the treatment. Adverse effects, adherence to therapy and patients' satisfaction were measured.

Clinical and histological parameters of photoaging were studied at baseline and after treatment. After completion of treatment with imiquimod, the final clinical evaluation was compared to the initial one.

DETAILED DESCRIPTION:
An experimental study was conducted between July and November 2010 in order to evaluate the efficacy and safety of imiquimod as a treatment option for photoaging.

The sample population was made up of individuals from both genders, older than 40 years, who worked at a flower growing farm located in a rural area of Rionegro (Antioquia) with an altitude of 2,125 meters above sea level; approximately composed of 80 people.

The sample size was calculated considering improvements in 50% or more of patients had to be detected, with a confidence interval of 95%, a power of 80%, a sampling error of 5%.

There were five visits: one at baseline and at months 1, 2, 3 and 4. In each visit patients were assesed clinically, a photograph was taken and adherence and side effects were investigated. Treatment was given during the first 3 months. A biopsy was taken at baseline and during the 4th month assessment. The last visit for clinical monitoring, photographic follow up and skin biopsy was at 16 weeks (4 weeks after discontinuation of the medication). In this last visit patient's satisfaction was evaluated through a survey.

The clinical assessment of photodamage performed by two dermatologists independently included: Changes in texture: dryness/roughness; changes in color: mottled hyperpigmentation, lentigines, yellowing; wrinkles: fine, deep wrinkles and laxity; telangiectasias.

Clinical signs like dryness, burning, erythema, itching, fissures and scabs were used to measure skin irritation.

Severity for the parameters measured in the clinical assessment of photoaging and the assessment of skin irritation was graded on a point scale of 0-3 where 0 was absence, one was mild, 2 moderate and 3 severe.

Biopsies were taken from sites adjacent to the temporal facial area. Aseptic iodine solution was used on the selected area, then the biopsy site was infiltrated with lidocaine 2% (about 0.5 cc) with a short 30-gauge needle and once analgesia was obtained a punch biopsy number 4 mm was taken. The skin biopsy was kept in a jar with formalin properly labeled and sent for histopathology. Then the biopsy site was sutured with 5-0 prolene. The biopsies were sent to the pathology department of the CES University for hematoxylin-eosin staining and they were blind - read by two dermatopathologists who evaluated the following parameters: epidermal changes: epidermal thickness, thickness of the granular layer, melanin content, atypia of melanocytes and keratinocytes, dermal-epidermal junction: pigment incontinence; dermis: inflammation, solar elastosis, fibrosis in the papillary dermis and telangiectasia.

Adherence was measured by asking patients in each one of the visits and it was considered excellent when the drug was applied 3 times per week, regular if the patient missed 2-3 applications between visits and poor if he/she missed more than 5 applications.

ELIGIBILITY:
Inclusion Criteria:

* patients with Fitzpatrick's skin types I to IV, with a photoaging equal to or greater than 3 on the Glogau measuring scale, who had not used systemic retinoids for over four weeks during six months prior to baseline,
* Patients nor had they undergone chemical peels or used exfoliants or applied botulinum toxin or any other abrasive substance on the face six months prior baseline
* patients that had not used topical retinoids or steroids two months prior to baseline
* patients that had not undergone facial rejuvenation surgery 12 months prior to treatment.

Exclusion Criteria:

* pregnant or nursing women
* patients currently being treated with phototherapy
* patients currently being treated with photochemotherapy or whom were scheduled to start
* patients with suspected skin cancer assessed by clinical examination
* patients with dermatological conditions with changes in the texture or color of the skin
* Patients with inflammatory dermatoses, immunological, infectious, or neoplastic skin diseases located in the periocular area since it could interfere with the clinical assessment of photoaging.
* Patients that at the time of inclusion expressed treatment refusal, disinterest or inability to comply with the protocol as well as those with skin types V and VI were not included.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinical response by percentage of improvement | 8 weeks
  To determine the degree of patient improvement percentages were set according to the values obtained in the first and last measurement as follows:
  For ordinal clinical variables that had 4 categories the following percentages were established: Slight 1-point improvement (1-32%), moderate 2-point improvement (33-66%), good 3-point improvement (> 66%), same or worse, one or more points of deterioration (<= 0%).
  For ordinal histological variables that were 4 categories the calculated improvement percentages were equal to the ones just described and for those with 5 variables, the established percentages were as follows: Slight 1-point improvement (1-25%), moderate 2-point improvement (26-50%), good 3-point improvement (51-75%), excellent 4-point improvement (> 75%), one or more points of deterioration (<= 0%).

CONTACTS AND LOCATIONS:
Overall Officials: Sol Beatriz Jiménez, MD, Study Director — CES University; Lucía Salinas, MD, Principal Investigator — CES University; Ana Cristina Ruíz, MD, Principal Investigator — CES University; Natalia De la Calle, MD, Principal Investigator — CES University; María Alejandra Zuluaga, MD, Principal Investigator — CES University; Rubén Darío Manrique, PhC, Principal Investigator — CES University; Bibiana Castro, MSc, Principal Investigator — CES University
Locations (1):
- Centro de servicios CES Sabaneta, Medellín, Antioquia, Colombia

REFERENCES:
- [Background] Giacomoni PU, Declercq L, Hellemans L, Maes D. Aging of human skin: review of a mechanistic model and first experimental data. IUBMB Life. 2000 Apr;49(4):259-63. doi: 10.1080/15216540050033104. PMID 10995026
- [Background] Glogau RG. Physiologic and structural changes associated with aging skin. Dermatol Clin. 1997 Oct;15(4):555-9. doi: 10.1016/s0733-8635(05)70465-4. PMID 9348456
- [Background] Fisher GJ, Wang ZQ, Datta SC, Varani J, Kang S, Voorhees JJ. Pathophysiology of premature skin aging induced by ultraviolet light. N Engl J Med. 1997 Nov 13;337(20):1419-28. doi: 10.1056/NEJM199711133372003. PMID 9358139
- [Background] Quan T, He T, Kang S, Voorhees JJ, Fisher GJ. Solar ultraviolet irradiation reduces collagen in photoaged human skin by blocking transforming growth factor-beta type II receptor/Smad signaling. Am J Pathol. 2004 Sep;165(3):741-51. doi: 10.1016/s0002-9440(10)63337-8. PMID 15331399
- [Background] Fisher GJ, Talwar HS, Lin J, Voorhees JJ. Molecular mechanisms of photoaging in human skin in vivo and their prevention by all-trans retinoic acid. Photochem Photobiol. 1999 Feb;69(2):154-7. doi: 10.1562/0031-8655(1999)0692.3.co;2. PMID 10048311
- [Background] Rabe JH, Mamelak AJ, McElgunn PJ, Morison WL, Sauder DN. Photoaging: mechanisms and repair. J Am Acad Dermatol. 2006 Jul;55(1):1-19. doi: 10.1016/j.jaad.2005.05.010. PMID 16781287
- [Background] Metcalf S, Crowson AN, Naylor M, Haque R, Cornelison R. Imiquimod as an antiaging agent. J Am Acad Dermatol. 2007 Mar;56(3):422-5. doi: 10.1016/j.jaad.2006.10.034. Epub 2006 Dec 20. PMID 17184874
- [Background] Ohnishi Y, Tajima S, Akiyama M, Ishibashi A, Kobayashi R, Horii I. Expression of elastin-related proteins and matrix metalloproteinases in actinic elastosis of sun-damaged skin. Arch Dermatol Res. 2000 Jan;292(1):27-31. doi: 10.1007/pl00007457. PMID 10664012
- [Background] Weinstein GD, Nigra TP, Pochi PE, Savin RC, Allan A, Benik K, Jeffes E, Lufrano L, Thorne EG. Topical tretinoin for treatment of photodamaged skin. A multicenter study. Arch Dermatol. 1991 May;127(5):659-65. PMID 2024983
- [Background] Kang SS, Kauls LS, Gaspari AA. Toll-like receptors: applications to dermatologic disease. J Am Acad Dermatol. 2006 Jun;54(6):951-83; quiz 983-6. doi: 10.1016/j.jaad.2005.05.004. PMID 16713451
- [Background] Dockrell DH, Kinghorn GR. Imiquimod and resiquimod as novel immunomodulators. J Antimicrob Chemother. 2001 Dec;48(6):751-5. doi: 10.1093/jac/48.6.751. PMID 11733457
- [Background] Sauder DN, Mofid MZ. Topical immunotherapy: what's new. Dermatol Clin. 2005 Apr;23(2):245-58. doi: 10.1016/j.det.2004.08.002. PMID 15837154
- [Background] Schon M, Schon MP. The antitumoral mode of action of imiquimod and other imidazoquinolines. Curr Med Chem. 2007;14(6):681-7. doi: 10.2174/092986707780059625. PMID 17346155
- [Background] Torres A, Storey L, Anders M, Miller RL, Bulbulian BJ, Jin J, Raghavan S, Lee J, Slade HB, Birmachu W. Immune-mediated changes in actinic keratosis following topical treatment with imiquimod 5% cream. J Transl Med. 2007 Jan 26;5:7. doi: 10.1186/1479-5876-5-7. PMID 17257431
- [Background] McInturff JE, Modlin RL, Kim J. The role of toll-like receptors in the pathogenesis and treatment of dermatological disease. J Invest Dermatol. 2005 Jul;125(1):1-8. doi: 10.1111/j.0022-202X.2004.23459.x. PMID 15982296
- [Background] Jobanputra KS, Rajpal AV, Nagpur NG. Imiquimod. Indian J Dermatol Venereol Leprol. 2006 Nov-Dec;72(6):466-9. doi: 10.4103/0378-6323.29352. No abstract available. PMID 17179631
- [Background] Smith K, Hamza S, Germain M, Skelton H. Does imiquimod histologically rejuvenate ultraviolet radiation-damaged skin? Dermatol Surg. 2007 Dec;33(12):1419-28; discussion 1428-9. doi: 10.1111/j.1524-4725.2007.33311.x. PMID 18076606
- [Background] Szeimies RM, Gerritsen MJ, Gupta G, Ortonne JP, Serresi S, Bichel J, Lee JH, Fox TL, Alomar A. Imiquimod 5% cream for the treatment of actinic keratosis: results from a phase III, randomized, double-blind, vehicle-controlled, clinical trial with histology. J Am Acad Dermatol. 2004 Oct;51(4):547-55. doi: 10.1016/j.jaad.2004.02.022. PMID 15389189
- [Result] Berneburg M, Plettenberg H, Krutmann J. Photoaging of human skin. Photodermatol Photoimmunol Photomed. 2000 Dec;16(6):239-44. doi: 10.1034/j.1600-0781.2000.160601.x. PMID 11132125